CLINICAL TRIAL: NCT03344835
Title: A Comprehensive Assessment of the Physical and Biological Effects of Patients With Prostate Cancer in Hong Kong
Brief Title: Hong Kong Prostate Cancer Study Group Database
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, NG Chi Fai, Professor NG, Chi Fai, Chinese University of Hong Kong
Other Study IDs: HK-CaP
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Disease Outcome
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prostate Cancer: Patients diagnosed with prostate cancer
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Prostate cancer (PCa) is ranked 3rd in annual incidence of male cancer and ranked 5th for cancer-related death in men in Hong Kong which accounts for about 9.1 deaths per 100,000 men in 2011. Its incidence is rising rapidly, almost tripled in the past 10 years. In Hong Kong, the two main screening methods for PCa are digital rectal examination (DRE) and serum prostate-specific antigen (PSA) level blood test, and the gold standard of diagnosis of PCa is transrectal ultrasound (TRUS) with prostate biopsy.

For those who diagnosed with PCa, there are different kinds of managements depending on patient's age group and disease stage. Watchful waiting is for older patients who presents with low-risk prostate cancer. And active surveillance is applicable to patients who are eligible for potentially curative management. While radiotherapy or radical prostatectomy are recommended as curative management for early stage PCa, androgen deprivation therapy (ADT) is the main treatment modality for advanced or recurrent prostate cancer. Advanced prostate cancer that recurrence is called castration refractory prostate cancer (CRPC). There are many new agents, including second line hormonal therapy, chemotherapy, androgen biosynthesis inhibitors, immunotherapy, bone targeting agents etc., available for the further management.

In this study, investigators would like to establish a local prostate cancer registry to facilitate the collection of clinical information and outcomes of prostate cancer management. Hopefully, this registry can provide information regarding the epidemiology, natural history, and treatment outcomes of local prostate cancer. The information would be helpful for research, public education, health care planning and also international collaboration. Ultimately, patients and public would be benefited from these works.

DETAILED DESCRIPTION:
The prostate gland is a clinically important male accessory sex gland and vital for its production of semen. Prostate cancer (PCa) is ranked 3rd in annual incidence of male cancer and ranked 5th for cancer-related death in men in Hong Kong which accounts for about 9.1 deaths per 100,000 men in 2011. Its incidence is rising rapidly, almost tripled in the past 10 years. Although this cancer is extremely rare before age 40 but the incidence increases with age, as the elderly population continues to increase, the impact of PCa on the men's health and also the burden on health care system will continue to rise. In addition to age, epidemiological data shows that race is also an important risk factor for prostate cancer. African-American men have the highest rates of prostate cancer in the world. For Asian populations, native Chinese and Japanese showed the lowest prostate cancer rates, though the incidence is rapidly increasing in the past decades.

The two main screening methods for PCa are digital rectal examination (DRE) and serum prostate-specific antigen (PSA) level blood test. DRE is an exam to check for growths or enlargement of the prostate gland. A tumor in the prostate can often be felt as a hard nodule. This may be done as a regular exam or check for the symptoms. If problems are suspected, DRE is usually done together with PSA, which was first introduced to evaluate the possibility of present of PCa in 1987. A common PSA threshold for biopsy in Hong Kong and Asia is PSA level greater than 4.0 ng/mL. Despite the controversial of PSA and some newer markers for PSA diagnosis, it is still the most common screening for PCa, due to the low cost and simplicity.

The gold standard of diagnosis of PCa is transrectal ultrasound (TRUS) with prostate biopsy. During the procedure, usually ten cores of biopsies will be taken and sent for pathological evaluation. If any of the biopsies are found malignant, Gleason score will be given and the stage of cancer will be determined.

Unlike other malignancy, PCa is characterized by its slow progression nature and even for metastatic disease the 5-year survival is up to 20%. Therefore, there will be different kinds of management for difference age group and disease stage: active surveillance (AS), watchful waiting, and treatments. Watchful waiting is for older patients who presents with low-risk prostate cancer. In these cases, treatment is probably not suitable for them due to the old age and low effectiveness. Contrasting watchful waiting, AS is applicable to patients who are eligible for potentially curative management. During AS, PCa is closely monitored for signs of progression. PSA blood test and DRE are usually administered at times along with a repeat biopsy of the prostate at one year and then at specific intervals thereafter. If symptoms develop, or if tests indicate the cancer is growing, treatment will be necessary.

For early stage of prostate cancer, radiotherapy or radical prostatectomy are recommended as curative management. The purpose of these treatments is to cure the disease. Over 80% of patients were cured with no recurrence. Currently, robotic prostatectomy is the main surgical approach for localized prostate cancer with acceptable perioperative results. Radiotherapy, both external beam and brachytherapy, are also standard therapy for prostate cancer. The overall complication rate, as reported from the Western literatures, for both surgery and radiotherapy are quite low. The final choice of treatment will largely depend on the join decision between physicians and patients.

However, for advanced or recurrent prostate cancer, androgen deprivation therapy (ADT) is the main treatment modality. While the effectiveness of ADT is well documented in the literature, the adverse effect profile in Asian patients, in particular to the cardiovascular system and bone metabolism, was not well documented.

Due to the continue changes in the behavior of prostate cancer cell under androgen deprivated environment, advanced prostate cancer will eventually entered a stage of castration refractory prostate cancer (CRPC). Currently, there are many new agents, including second line hormonal therapy, chemotherapy, androgen biosynthesis inhibitors, immunotherapy, bone targeting agents etc., available for the further management of these CRPC patients. Unfortunately, the clinical outcome and side effect profiles for further treatment for patients with in local Chinese population, as well as in Asian population was still not that certain.

Due to the continue changes in the behavior of prostate cancer cell under androgen deprived environment, advanced prostate cancer will eventually entered a stage of castration refractory prostate cancer (CRPC). Currently, there are many new agents, including second line hormonal therapy, chemotherapy, androgen biosynthesis inhibitors, immunotherapy, bone targeting agents etc., available for the further management of these CRPC patients. Unfortunately, the clinical outcome and side effect profiles for further treatment for patients with in local Chinese population, as well as in Asian population was still not that certain.

Facing the increase in clinical demand by the drastic increase in patient population, together with the rapid development in various therapies for different stages of prostate cancer, there is a need to have better understanding about the natural history, clinical outcomes of various therapies for prostate cancer. Therefore, investigators would like to establish a local prostate cancer registry to facilitate the collection of clinical information and outcomes of prostate cancer management. Hopefully, this registry can provide information regarding the epidemiology, natural history, and treatment outcomes of local prostate cancer. The information would be helpful for research, public education, health care planning and also international collaboration. Ultimately, patients and public would be benefited from these works

In this study, both retrospective and prospective cohort study design will be adopted. Patients diagnosed with prostate cancer from 2016 will be captured prospectively and those who diagnosed in or before 2015 will be captured retrospectively. Patients diagnosed with prostate cancer in the hospitals under the New Territories East Cluster (NTEC) & New Territories West Cluster (NTWC) will be identified in specialist clinics, wards, and during TRUS, and then enrolled to the study. This study will be conducted by observation; no intervention article is used. The time of diagnosis of prostate cancer will be set as baseline of that subject. All the demographic and medical background will be traced back. All patients will be followed up every 6 months and thereafter. During the follow-up, patients' medical status including survival, cancer status, treatment, complications will be captured from the medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the age of 18 or above
* Patients with clinical diagnosis of prostate cancer

Exclusion Criteria:

* Patients diagnosed to have ductal type of prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer only happens in male patients
Study Population: All patients diagnosed with prostate cancer, in NDH, PWH and TMH, since 1995 would be included in the registry. Both retrospective and prospective cohort study design will be adopted in this study. Patients diagnosed with prostate cancer in the hospitals under the NTEC & NTWC cluster will be identified in specialist clinics, wards, and during TRUS, and then enrolled to the study.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Specific survival | 10 years
  The cancer specific survival of different disease stages in Hong Kong Chinese prostate cancer patients

SECONDARY OUTCOMES:
Overall survival | 10 years
  Overall Survival of different disease stages in Hong Kong Chinese prostate cancer patients
Biological progress | 10 years
  Time to biochemical progression of different disease stages in Hong Kong Chinese prostate cancer patients
PSA response | 10 years
  PSA response for different treatment modalities at different disease stages
Complications rate | 10 years
  Complications rate of different modalities of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiu PK, Wong AY, Hou SM, Yip SK, Ng CF. Effect of body mass index on serum prostate-specific antigen levels among patients presenting with lower urinary tract symptoms. Asian Pac J Cancer Prev. 2011;12(8):1937-40. PMID 22292628
- [Background] Ng CF, Chiu PK, Lam NY, Lam HC, Lee KW, Hou SS. The Prostate Health Index in predicting initial prostate biopsy outcomes in Asian men with prostate-specific antigen levels of 4-10 ng/mL. Int Urol Nephrol. 2014 Apr;46(4):711-7. doi: 10.1007/s11255-013-0582-0. Epub 2013 Oct 18. PMID 24136184
- [Background] Sasagawa I, Nakada T. Epidemiology of prostatic cancer in East Asia. Arch Androl. 2001 Nov-Dec;47(3):195-201. doi: 10.1080/014850101753145906. PMID 11695843
- [Background] Ng CF, Yeung R, Chiu PK, Lam NY, Chow J, Chan B. The role of urine prostate cancer antigen 3 mRNA levels in the diagnosis of prostate cancer among Hong Kong Chinese patients. Hong Kong Med J. 2012 Dec;18(6):459-65. PMID 23223645
- [Background] Sim HG, Cheng CW. Changing demography of prostate cancer in Asia. Eur J Cancer. 2005 Apr;41(6):834-45. doi: 10.1016/j.ejca.2004.12.033. PMID 15808953
- [Background] Wang W, Yuasa T, Tsuchiya N, Maita S, Kumazawa T, Inoue T, Saito M, Ma Z, Obara T, Tsuruta H, Satoh S, Habuchi T. Bone mineral density in Japanese prostate cancer patients under androgen-deprivation therapy. Endocr Relat Cancer. 2008 Dec;15(4):943-52. doi: 10.1677/ERC-08-0116. Epub 2008 Jul 30. PMID 18667685
- [Background] Wilt TJ, Thompson IM. Clinically localised prostate cancer. BMJ. 2006 Nov 25;333(7578):1102-6. doi: 10.1136/bmj.39022.423588.DE. No abstract available. PMID 17124221
- [Background] Wilt TJ, MacDonald R, Rutks I, Shamliyan TA, Taylor BC, Kane RL. Systematic review: comparative effectiveness and harms of treatments for clinically localized prostate cancer. Ann Intern Med. 2008 Mar 18;148(6):435-48. doi: 10.7326/0003-4819-148-6-200803180-00209. Epub 2008 Feb 4. PMID 18252677
- [Background] Yip KH, Yee CH, Ng CF, Lam NY, Ho KL, Ma WK, Li CM, Hou SM, Tam PC, Yiu MK, Fan CW. Robot-assisted radical prostatectomy in Hong Kong: a review of 235 cases. J Endourol. 2012 Mar;26(3):258-63. doi: 10.1089/end.2011.0303. Epub 2012 Jan 4. PMID 22192108